CLINICAL TRIAL: NCT06202196
Title: Evaluate the Impact of a Specific Risk Prevention Program Associated With a Therapeutic Patient Education Program on the Risk Behaviors of Adult Patients With Uncontrolled Epilepsy.
Brief Title: Risk Prevention Program and Therapeutic Patient Education Program of Patients With Uncontrolled Epilepsy
Acronym: EPI-RISK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL18_0196
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; Therapeutic Patient Education
MeSH Terms: conditions — Epilepsy | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This clinical study is a multicenter, open-label, randomized in two parallel groups of patients: an experimental group "specific plan for the prevention of risks related to epilepsy" and a control group "usual consultations with the neurologist and the usual TPE sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients of the experimental group will have therapeutic patient education sessions that include one "Recognizing and Managing the Risks of Epilepsy" workshop.
  Interventions: Procedure: Risk prevention session
- Control group "Usual management" (Other): Patients of the "control" group will have the usual therapeutic patient education sessions.
  Interventions: Procedure: Usual Therapeutic Patient Education (TPE) management

INTERVENTIONS:
Procedure: Risk prevention session — The patient will have a consultation dedicated to information on the risks with the neurologist within 1 to 3 months (during this period, the patient must complete the seizure diary).
  An appointment with the psychologist within 2 weeks +/- 1 week following the risk discussion consultation will also be scheduled. In this interval of 2 weeks, the patient will have the possibility of reaching the neurologist, the psychologist or the nurse by telephone if he feels the need.
  Then participants will be proposed the therapeutic education session including a workshop called ""Recognizing and Managing the Risks of Epilepsy". The last visit 3 months after the last session will assess differents questionnaires/scales including the Epilepsy Self Management Scale (ESMS).
  Arms: Experimental group
Procedure: Usual Therapeutic Patient Education (TPE) management — The control group will have usual follow-up including consultations with the neurologist and follow-up of the usual TPE program, namely the individual interview and follow-up of the usual TPE workshops for each center.
  Arms: Control group "Usual management"

SUMMARY:
Pilot, controled, randomized study aiming to evaluate a plan for the prevention of risks related to epilepsy, 3 months after the last therapeutic patient education session. Two groups of patients will be compared: group "intervention" (consultation with the neurologist then a psychologist followed by a session dedicated to risk prevention ("Recognize and Manage risks") integrated into usual Therapeutic Patient Education (TPE) versus "control" group (usual consultations with the neurologist and usual TPE).

37 subjects per group will be included in this study.

DETAILED DESCRIPTION:
The study will be proposed to patients with uncontrolled epilepsy (n=74) aged 18 to 40.

The investigators will evaluate 3 months after the last therapeutic patient session, the impact of the epilepsy-related risk prevention system on the self-management of epilepsy ("Safety Management" score of the Epilepsy Self Management Scale (ESMS). This scale has 5 dimensions (5 sub-scores): treatment management, information management, safety management, seizure management and lifestyle management.

Each clinical investigation team works in collaboration with a clinical psychologist for psychological assessment interviews.

The implementation of such a plan should enable patient to acquire so-called safety skills aimed at protecting his life, reducing risky behavior and increasing medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years old
* Patient with poorly controlled epilepsy (persistence of seizures evolving for more than a year despite proper treatment) or patient seizure-free for over a year but for whom therapeutic patient education (TPE) would be beneficial according to the investigator..
* Patient agreeing to participate in a therapeutic education program (TPE)

Exclusion Criteria:

* Epileptic patient who has already benefited from a TPE epilepsy program
* Patients with major cognitive impairment
* Patient under guardianship or legal protection (safeguard of justice)
* Pregnant or breast-feeding women
* Failure to obtain written informed consent after a reflection period
* Patient who for geographical, social or psychological reasons could not participate in the research
* Any situation that, in the opinion of the investigator, could present risks to the patient and to the research
* Participation in another therapeutic research
* Subjects not covered by public health insurance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2028-04-16 (Estimated); Study Completion 2028-04-16 (Estimated)

PRIMARY OUTCOMES:
Change in the "safety management" sub-scale of the Epilepsy Self Management Scale (ESMS) | From baseline to 3 months after the end of TPE
  The ESMS is a 38-item scale that assesses the frequency of use of self-management strategies in epilepsy. This scale has 5 dimensions (5 sub-scores):management of treatments, information, safety, epileptic seizures and lifestyle.
  Each item can be rated from 1 (never) to 5 (always) depending on the frequency of use of self-management strategies.

SECONDARY OUTCOMES:
Global score of Epilepsy Self Management Scale (ESMS) | From baseline to 3 months after the end of TPE
  The total possible scores of the ESMS range from 38 to 190 with higher scores indicating greater use of self-management strategies.
Sub-scales of Epilepsy Self Management Scale (ESMS) | From baseline to 3 months after the end of TPE
  The following subscales will be calculated : realms of medication management (10 items), information management (8 items), seizure management (6 items), and lifestyle management (6 items).
Medication adherence rating scale "MARS" | From baseline to 3 months after the end of TPE
  The measurement of compliance will be based on the MARS scale (medication adherence rating scale) composed of 10 items. This questionnaire is one of the most widely used, particularly in the field of neuropsychiatry. This scale does not have a threshold. Items 1 to 4 correspond to treatment adherence behavior, items 5 to 8 correspond to attitude around drug intake and items 9 and 10 are reversed: negative effect of treatments and attitude towards the psychotropic drug.
Scores on the Generalized Anxiety Disorders Scale (GAD-7) | From baseline to 3 months after the end of TPE
  Scores on the Generalized Anxiety Disorders Scale (GAD-7). The GAD-7 is a self-administered questionnaire consisting of 7 items rated from 0 to 3. The total score is obtained by adding the score obtained for each item (score ranging from 0 to 21). A total score strictly greater than 7 should raise suspicion of a generalized anxiety disorder.
Neurological Disorders Depression Inventory for Epilepsie (NDDI-E) Score | From baseline to 3 months after the end of TPE
  The NDDI-E is a scale validated in French for screening major depressive episodes (characterized) in patients with epilepsy. This is a self-administered questionnaire (completed by the patient). The total score is obtained by adding the score obtained at each item. A total score strictly greater than 15 should raise suspicion of a major depressive episode. The NDDI-E is a screening scale. If the score is > 15, it is therefore advisable to have the diagnosis confirmed by a clinical psychiatric assessment.
Quality of Life in Epilepsy Inventory (QOLIE-31) score | From baseline to 3 months after the end of TPE
  QOLIE-31 (validated French version) is an epilepsy-related quality of life scale that includes 31 items on health and daily activities (Cramer et al., 1998).
  The QOLIE-31 contains seven multi-item scales that tap the following healths concepts: emotional well-being, social functioning, energy/fatigue, cognitive functioning, seizure worry, medication effects and overall quality of life. A QOLIE-31 overall score is obtained using a weighted average of the multi-item scale scores.
Questionnaire on "knowledge and assessment of risky behaviors" | From baseline to 3 months after the end of TPE
  Questionnaire on "knowledge and assessment of risky behaviors" (i.e driving, risky sports, alcohol intake, sleep deprivation, bathing, swimming, burns)
Frequency of seizures | From baseline to 3 months after the end of TPE
  Frequency of seizures will be recorded on a patient diary
Seizures description | From baseline to 3 months after the end of TPE
  Seizures decription will be recorded on a patient diary

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Gui de Chauliac, Montpellier, France